CLINICAL TRIAL: NCT04328675
Title: Registration Study of Natural History and Clinical Characteristics of Amyotrophic Lateral Sclerosis (ALS) in Mainland China
Brief Title: Registration Study of Amyotrophic Lateral Sclerosis (ALS) in Mainland China
Acronym: ChALSR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FDongsheng-81873784
Record Dates: First submitted 2020-03-17; First posted 2020-03-31 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-03

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A multi-center registration study of natural history and clinical characteristics of ALS in mainland China

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a rapidly progressive neurodegenerative disease of unknown etiology that is currently incurable. This study is a national multi-center registration study. The study collects general information of ALS patients including medical history, disease characteristics, clinical treatment data, and patient information for different visits in different centers. The aim of the study is: a) describe the distribution of ALS in mainland China(explore the differences in the number of ALS at different times, different regions, and different populations) and further find the reasons that affect the distribution of ALS, b) study the development of ALS in mainland China and the corresponding changes in the characteristics of the disease, c) explore factors that influence the prognosis of ALS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of laboratory-supported probable, probable, or definite ALS according to EI Escorial diagnostic criteria
* Age: 18-70 years

Exclusion Criteria:

* Refuse to cooperate or reject the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the criteria will be enrolled from multi-centers in mainland China.
Sampling Method: Non-Probability Sample
Enrollment: 4752 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2023-03-20 (Estimated); Study Completion 2023-03-20 (Estimated)

PRIMARY OUTCOMES:
Effective Survival | through study completion, an average of 3 month
  The length of time from the date of diagnosis to patient death or tracheotomy or ventilator-assisted breathing.

SECONDARY OUTCOMES:
Overall Survival | through study completion, an average of 3 month
  The length of time from the date of diagnosis to patient death due to any cause or the last confirmed survival.
Rate of disease progression | through study completion, an average of 3 month
  The slope of decline of the ALS Functional Rating Scale-Revised (ALSFRS-R) score from the diagnosis time to the follow-up time. ALSFRS-R values from 0 to 48 and it implies better outcome when it is higher.
Rate of Weight decline | through study completion, an average of 3 month
  The slope of decline of weight
Rate of BMI decline | through study completion, an average of 3 month
  The slope of decline of BMI
Rate of Forced Vital Capacity (FVC) | through study completion, an average of 3 month
  The slope of decline of Forced Vital Capacity (FVC) to assess the respiratory function.

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, MD, PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] He J, Fu JY, Chen L, He J, Dang J, Zou Z, Ma S, Li N, Fan D. Multicentre, prospective registry study of amyotrophic lateral sclerosis in mainland China (CHALSR): study protocol. BMJ Open. 2020 Dec 4;10(12):e042603. doi: 10.1136/bmjopen-2020-042603. PMID 33277290